CLINICAL TRIAL: NCT02109887
Title: Assessment of CMV-specific ELISPOT Assay for Predicting CMV Co-infection in Patients With Pneumocystitis Pneumonia (ACE-PCP)
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Associate Professor, Asan Medical Center
Other Study IDs: S2013-1999-0005; 2014-0198 (Other: Asan Medical Center)
Record Dates: First submitted 2014-03-31; First posted 2014-04-10 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Non-HIV Patients With Pneumocystis Jiroveci Pneumonia
Keywords: Pneumocystis jiroveci, cytomegalovirus, co-infection
MeSH Terms: conditions — Coinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PCP with true CMV co-infection
- PCP with innocent bystander CMV
- PCP without any evidence of CMV

SUMMARY:
PCP (Pneumocystis jiroveci pneumonia) is one of the important opportunistic infections in immunocompromised patients including HIV-infected patients, transplant recipients, and immunosuppressant users. About one third of non-HIV patients with PCP have the evidence of co-infection with CMV. In this difficult clinical situation, physicians have difficulty to decide on whether anti-CMV treament will help patients with any evidence of CMV co-infection. However, there is no objective test to differentiate true co-infection of CMV from innocent bystander of CMV in those with PCP. The investigators thus evaluate the usefulness of CMV-specific ELISPOT assay in patients with PCP to differentiate true co-infection of CMV from inocent bystander of CMV. This findings may guide physicians to decide anti-CMV treatment in patients with PCP and CMV co-infection.

DETAILED DESCRIPTION:
PCP (Pneumocystis jiroveci pneumonia) is one of the important opportunistic infections in immunocompromised patients including HIV-infected patients, transplant recipients, and immunosuppressant users. About one third of non-HIV patients with PCP have the evidence of co-infection with CMV. In this difficult clinical situation, physicians have difficulty to decide on whether anti-CMV treament will help patients with any evidence of CMV co-infection. However, there is no objective test to differentiate true co-infection of CMV from innocent bystander of CMV in those with PCP. The investigators thus evaluate the usefulness of CMV-specific ELISPOT assay in patients with PCP to differentiate true co-infection of CMV from inocent bystander of CMV. This findings may guide physicians to decide anti-CMV treatment in patients with PCP and CMV co-infection.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PCP based on PCP immunohistochemistry or PCP PCR
* age 16 or more
* agree with written informed consent
* WBC count 2000/uL or more

Exclusion Criteria:

* HIV infection

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-HIV patients with PCP
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
CMV co-infection | 1 month after the diagnosis of PCP
  CMV co-infection is defined as (1) positive BAL (bronchoalveolar lavage fluid) CMV culture and (2) ganciclovir therapy for at least 1 week.

SECONDARY OUTCOMES:
overall mortality | 1 month after the diagnosis of PCP
innocent bystander CMV infection | 1 month after the diagnosis of PCP
  innocent bystander CMV infection
  * positive blood CMV antigenemia and/or positive blood or BAL CMV qPCR without positive BAL CMV culture
  * clinical improvement without ganciclovir therapy for at least 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea